CLINICAL TRIAL: NCT07057440
Title: Effect of Nicotine Pouches on The Underlying Normal Electrocardiogram A Double-Blinded, Placebo-Controlled Cross-over Study Exploring the Dose-Response Effects of Nicotine Pouches on Heart Rate and the Electrocardiogram ACRONYM: The NICOTUNE Study
Brief Title: Effect of Nicotine Pouches on The Underlying Normal Electrocardiogram
Acronym: NICOTUNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ekim Seven (Other)
Responsible Party: Sponsor-Investigator, Ekim Seven, Cardiologist, PhD, clinical associate professor, department of cardiology, Hvidovre University Hospital, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-25018523
Record Dates: First submitted 2025-06-10; First posted 2025-07-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Heart Rate; ECG; Vital Sign Monitoring; Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo pouch arm (Placebo Comparator)
  Interventions: Other: Placebo Pouch
- Low-dosage nicotine pouch arm (Experimental)
  Interventions: Other: Low Dose Nicotine Pouch
- High-dosage nicotine pouch arm (Experimental)
  Interventions: Other: High-dose Nicotine Pouch

INTERVENTIONS:
Other: High-dose Nicotine Pouch — A High Dose Nicotine Pouch are placed and held in the oral cavity (between the gum and lip) for 20 minutes, as per standard use instructions.
  After 20 minutes pouches are removed from the oral cavity and disposed.
  Arms: High-dosage nicotine pouch arm
Other: Low Dose Nicotine Pouch — A Low Dose Nicotine Pouch are placed and held in the oral cavity (between the gum and lip) for 20 minutes, as per standard use instructions. After 20 minutes pouches are removed from the oral cavity and disposed.
  Arms: Low-dosage nicotine pouch arm
Other: Placebo Pouch — A Placebo Pouch are placed and held in the oral cavity (between the gum and lip) for 20 minutes, as per standard use instructions. After 20 minutes pouches are removed from the oral cavity and disposed.
  Arms: Placebo pouch arm

SUMMARY:
Nicotine pouches (NPs) are increasingly being used by children, adolescents, and adults, and are often presented as a less harmful alternative to, for example, smoking. The ability to use these products discreetly (unlike smoking) makes them an attractive option for individuals who wish to avoid the stigma that smokers may sometimes experience.

Nicotine is a well-known addictive substance that affects many organ systems, including the heart and circulatory system. The amount of nicotine in NPs varies greatly, but the pouches can contain large amounts of nicotine compared to the content of a single cigarette. While many studies have previously examined the effects of smoking and other nicotine products on the heart and circulatory system, specific data on the effects of NPs on these same systems are rather limited.

In light of the above, the investigators have planned a study to investigate whether NPs affect the circulatory system and heart rate, assessed through electrocardiography (ECG) and vital signs (i.e., pulse, blood pressure, respiratory rate, and more).

The investigators hypothesis is that the nicotine content in NPs leads to notable changes in the aforementioned measurements and could therefore potentially be associated with an increased health risk.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years.
* Regular (defined as daily) or occasional (generally defined as nondaily) nicotine users (e.g., cigarettes, vaping, or nicotine pouches).
* Willingness to abstain from nicotine, caffeine (including caffeine containing energy drinks), and alcohol for 6 hours prior to the session

Exclusion Criteria:

* History of cardiovascular conditions.
* Medications affecting cardiac conduction or autonomic function (e.g., antiarrhythmic drugs).
* Pregnancy or breastfeeding.
* Current illness or infection.
* History of substance abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Heart rate | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Changes in HR (beats/minute) obtained from an ECG recorded 20 minutes after nicotine pouch administration compared to the baseline ECG.

SECONDARY OUTCOMES:
ECG parameters | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Changes in various ECG parameters from baseline:
  • PR interval (msec)
  • QRS duration (msec)
  • QT interval (corrected, QTc) (msec)
  • HRV (msec)
ST-T segment changes | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  ST-T segment changes, e.g., depression/elevation/inversion (mm) from baseline
Arrhythmias | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Any arrhythmias e.g., ectopic beats (yes/no, numerical) detected on the ECG compared with baseline ECG

OTHER OUTCOMES:
Blood pressure | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Changes in Blood pressure (mmHg)
Respiratory rate | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Changes in Respiratory rate (breaths per minute)
Oxygen saturation | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Changes in Oxygen saturation (percentage/%)
Body temperature | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Changes in Body temperature (degree Celsius)
Self-reported symptoms | 10 and 20 minutes (just before disposal) after the placement of the nicotine pouch in the oral cavity
  Subjective symptoms self-reported by the participants during the intervention using VAS-questionnaire of 10 known nicotine effect/symptoms (nausea, dizziness, lightheadedness, nervousness, sweatiness, headache, excessive salivation, heart pounding, confusion, and weakness).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of cardiology, Copenhagen University Hospital, Amager & Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided